CLINICAL TRIAL: NCT07254195
Title: Intensive Motor Rehabilitation of Stroke Patients: Evaluation of a Telerehabilitation Program
Brief Title: Assessment of an Intensive Motor Telerehabilitation Program for Stroke Patients
Acronym: REACT-AVC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL24_0504; 2025-A01054-45 (Other: ID-RCB)
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Stroke
Keywords: Stroke; motor; telerehabilitation; intensive therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR1 (Other): Immediately following discharge from the rehabilitation unit, patients will participate in a 12-weeks telerehabilitation program using the MindMotion GO device, in parallel to the standard care.
  During the 12-weeks program, patients will aim to achieve at least 300 minutes of active therapy time per week using the MindMotion GO device at their home. They will have 1 synchronous rehabilitation session per week in clinic or remotely via videoconference with a PT or an OT. The rest of the sessions will be done asynchronously and independently by the patient. The activity schedule will be drawn up by a therapist remotely and will be personalized for each patient.
  After 12 weeks, the patients will be asked whether they wish to continue with the telerehabilitation program. Patients who agree to continue will pursue the program for another 12 weeks, in parallel to standard care.
  Patients who do not want to continue the program will only receive standard care for the following 12 weeks.
  Interventions: Device: Telerehabilitation program using the MindMotion GO device
- TR2 (Other): Following discharge from the rehabilitation unit, patients will receive only standard care for 12 weeks.
  Then, they will start the telerehabilitation program using the MindMotion GO device for 12 weeks, in parallel to the standard care. During the 12-weeks program, patients will aim to achieve at least 300 minutes of active therapy time per week using the MindMotion GO device at their home. They will have 1 synchronous rehabilitation session per week in clinic or remotely via videoconference with a PT or an OT. The rest of the sessions will be done asynchronously and independently by the patient. The activity schedule will be drawn up by a therapist remotely and will be personalized for each patient.
  Interventions: Device: Telerehabilitation program using the MindMotion GO device

INTERVENTIONS:
Device: Telerehabilitation program using the MindMotion GO device — In parallel to the standard of care, patients will participate in a 12-weeks telerehabilitation program using the MindMotion GO device.
  MindMotion GO is a digital therapy device that offers a catalog of interactive games designed specifically for patients with neurological injuries.
  During the telerehabilitation program, patients will aim to achieve at least 300 minutes of active therapy per week. They will have 1 synchronous session per week in the clinic or remotely by videoconference with a therapist (PT or OT). Patients are expected to carry out the other planned sessions independently at home. The activity schedule will be drawn up by a remote therapist each week and will be personalized for each patient.

SUMMARY:
Stroke is a major cause of motor disability, particularly hemiplegia, and its incidence is increasing as the population ages. Despite partial spontaneous recovery in the first three months, 80% of patients retain a motor deficit after six months, requiring intensive rehabilitation to maximize recovery. However, after hospitalization, access to intensive rehabilitation is limited, due to geographical and mobility constraints, and the lack of reimbursement for private occupational therapy.

Telerehabilitation, using digital technologies, can overcome these difficulties by offering interactive, accessible rehabilitation at home. Studies show that its effectiveness is comparable to that of clinical rehabilitation.

Our study therefore proposes to evaluate the feasibility and effects of a home-based telerehabilitation program using the MindMotion GO device (MindMaze). This 12-week program aims to provide an additional intensive dose of rehabilitation to the standard of care, with 300 minutes of weekly active therapy, planned and monitored remotely by a therapist.

DETAILED DESCRIPTION:
Stroke is a major cause of motor disability, particularly hemiplegia, and its incidence is increasing as the population ages. Despite partial spontaneous recovery in the first three months, 80% of patients retain a motor deficit after six months, requiring intensive rehabilitation to maximize recovery. However, after hospitalization, access to intensive rehabilitation is limited, due to geographical and mobility constraints, and the lack of reimbursement for private occupational therapy.

Telerehabilitation, using digital technologies, can overcome these difficulties by offering interactive, accessible rehabilitation at home. Studies show that its effectiveness is comparable to that of clinical rehabilitation.

Our study therefore proposes to evaluate the feasibility and effects of a home-based telerehabilitation program using the MindMotion GO device (MindMaze). This 12-week program aims to provide an additional intensive dose of rehabilitation to the standard of care, with 300 minutes of weekly active therapy, planned and monitored remotely by a therapist. It combines synchronous (1time a week with a therapist) and asynchronous (autonomous) sessions.

This program is integrated into the post-stroke care pathway by facilitating the transition from hospital to home, without prolonging hospitalization or increasing face-to-face sessions.

The study will be a single-center randomized controlled trial, targeting patients in the sub-acute and chronic stages of stroke.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for a first ischemic or hemorrhagic stroke
* Stroke occurrence more than 30 days prior
* Presenting motor deficits affecting the upper limb, with or without involvement of the lower limb
* Able to follow the instructions of the home program using the MindMotion GO device
* Having at home an accessible email address, an Internet connection with password, a smartphone, a screen or TV with HDMI input (Full HD 1080p resolution), and a free space of approximately 1 m x 2.5 m in front of the screen
* Ability to sit without assistance
* Patient agreeing to participate in the study by signing an informed consent form
* Affiliated with, or entitled to, a social security scheme

Exclusion Criteria:

History of stroke

* Neurological pathology other than stroke
* Patient with uncontrolled epilepsy or seizure disorder
* Cardiac disease limiting exercise
* Pain limiting rehabilitation dose
* Major comprehension problems or severe psychiatric and/or cognitive disorders that could compromise understanding of the protocol and the smooth running of the study.
* Uncorrected hearing or visual deficits
* Severe apraxia
* Severe memory impairment
* Severe unilateral spatial neglect
* Total plegia of affected limb
* Pregnant, parturient or breast-feeding women
* Persons deprived of their liberty by judicial or administrative decision
* Persons admitted to a health or social institution for purposes other than research
* Adults under legal protection (guardianship, curatorship)
* Subjects participating in other intervention research.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2027-10-25 (Estimated); Study Completion 2027-10-25 (Estimated)

PRIMARY OUTCOMES:
Variation in the Goal Attainment Scale (GAS) score. | Baseline, at 8, 20, 32 and 44 weeks
  The GAS is used to measure achievement of individual goals. GAS goals will be set for each participant before the start of the intervention. Achievement of each objective will be rated on a 5-point scale: -2 (patient's initial, pre-intervention level), -1 (progress towards goal, without complete attainment), 0 (expected level), +1 (goal achieved better than expected), +2 (best hoped-for result).

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Henry Gabrielle, Saint-Genis-Laval, Lyon, France